CLINICAL TRIAL: NCT00293670
Title: Intermittent Vs Continuous Androgen Deprivation in Patients With Advanced Prostate Cancer
Brief Title: FINNPROSTATE Study VII: Intermittent Versus Continuous Androgen Deprivation in Patients With Advanced Prostate Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tampere University (Other)
Collaborators: Finnish Prostate Cancer Group (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9393FN/0001
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2006-02-17 (Estimated); Status verified 2006-02

CONDITIONS: Patients With T1-4 Advanced Prostate Cancer
MeSH Terms: interventions — Goserelin

INTERVENTIONS:
Drug: Goserelin (Zoladex)

SUMMARY:
To compare intermittent androgen deprivation (LHRHa treatment) with continuous androgen deprivation (LHRHa treatment or orchidectomy)

ELIGIBILITY:
• Inclusion Criteria (run-in period): T1-T4, metastatic (M1) prostate cancer T1-T4, non-metastatic (M0) prostate cancer with PSA > 60 ng/mL T3-T4, non-metastatic (M0) prostate cancer with PSA > 20ng/mL T1-T4, N+ prostate cancer WHO performance status 0-2 Written informed consent

• Inclusion criteria to the randomised period: Patients who fulfilled all entry criteria of the run-in period Patients who completed the 24-week run-in period Patients who responded to the 24-week run-in period with a decrease of PSA to < 10 ng/mL. If the baseline was < 20ng/mL, at least 50% decrease from the baseline measurement is required

Exclusion Criteria (run-in period):

Any previous or concurrent treatment of prostate cancer, except TURP, 5-alpha reductase inhibitor, radical prostatectomy or radiotherapy Any medication/treatment affecting sex hormone status

-

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 573
Dates: Start 1997-05; Study Completion 2015-04

PRIMARY OUTCOMES:
Time To Progression (TTP)

SECONDARY OUTCOMES:
Overall and prostate cancer-specific survival, time to treatment failure, quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Teuvo L Tammela, Professor, Principal Investigator — Tampere University Central Hospital, Finland
Locations (1):
- TUCH (Tampere University Central Hospital), Tampere, Finland

REFERENCES:
- [Derived] Salonen AJ, Taari K, Ala-Opas M, Viitanen J, Lundstedt S, Tammela TL; FinnProstate Group. Advanced prostate cancer treated with intermittent or continuous androgen deprivation in the randomised FinnProstate Study VII: quality of life and adverse effects. Eur Urol. 2013 Jan;63(1):111-20. doi: 10.1016/j.eururo.2012.07.040. Epub 2012 Jul 27. PMID 22857983
- [Derived] Salonen AJ, Taari K, Ala-Opas M, Viitanen J, Lundstedt S, Tammela TL; FinnProstate Group. The FinnProstate Study VII: intermittent versus continuous androgen deprivation in patients with advanced prostate cancer. J Urol. 2012 Jun;187(6):2074-81. doi: 10.1016/j.juro.2012.01.122. Epub 2012 Apr 11. PMID 22498230